CLINICAL TRIAL: NCT07039682
Title: Developing a Digital-Based Education and Self-Screening Model to Improve Knowledge, Self-Awareness, and HIV Testing Coverage Among Adolescents
Brief Title: Empowering Knowledge, Self-Testing & Resilience Through Innovative Methods for HIV
Acronym: EKSTRIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Rizka Ayu Setyani, Universitas Sebelas Maret, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 63/UN27.06.11/KEP/EC/2025; 400422-409 (Other Grant/Funding Number: Foreign, Commonwealth & Development Office (FCDO), British Embassy Jakarta)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection; HIV Prevention; Adolescent Health; Digital Education Interventions; Digital Health Intervention; Health Education; HIV Stigma
Keywords: hiv prevention; adolescent health; health education; digital intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study uses a double-blind design in which both participants and investigators are unaware of group allocation (intervention or control). The outcomes assessor is also blinded to minimize assessment bias. Only the data analyst, independent from the implementation team, will have access to the allocation code after data collection is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital HIV Education and Self-Screening (EKSTRIM Model) (Experimental): Participants in this arm will receive access to the EKSTRIM platform, a web-based digital tool designed for adolescents. The platform includes interactive educational content on HIV prevention, a self-assessment screening tool to evaluate individual HIV risk, and online peer educator support. The intervention will be implemented over a 6-week period. Participants will be encouraged to use the platform independently, with monitoring of access logs and engagement levels.
  Interventions: Device: Digital HIV Education and Self-Screening (EKSTRIM Model)
- Standard/Usual HIV Education Program (No Intervention): Participants in this arm will receive standard HIV-related education as provided through the school health program. This includes printed materials and classroom-based health education without access to digital tools or peer educator interaction. This group will serve as the comparison to evaluate the added impact of the digital EKSTRIM intervention.

INTERVENTIONS:
Device: Digital HIV Education and Self-Screening (EKSTRIM Model) — Participants in this arm will receive access to the EKSTRIM platform, a web-based digital tool designed for adolescents. The platform includes interactive educational content on HIV prevention, a self-assessment screening tool to evaluate individual HIV risk, and online peer educator support. The intervention will be implemented over a 6-week period. Participants will be encouraged to use the platform independently, with monitoring of access logs and engagement levels.
  Arms: Digital HIV Education and Self-Screening (EKSTRIM Model)

SUMMARY:
The goal of this study is to learn whether a digital tool can help improve HIV knowledge, self-awareness, and testing among adolescents in Yogyakarta, Indonesia. The tool includes online HIV education, a self-assessment for HIV risk, and access to trained peer educators for support. The study will also explore how comfortable and willing adolescents are to use this kind of digital health service.

The main questions the study aims to answer are:

* Can this digital tool help adolescents better understand HIV and their personal risk?
* Will more adolescents be willing to get tested for HIV after using the tool?
* What factors affect whether adolescents accept and use digital HIV services?

Researchers will compare two groups of high school students:

* One group will use the digital tool for 6 weeks
* The other group will receive standard HIV education (not through the tool)

Participants will:

* Answer surveys before and after the 6-week period
* Learn about HIV through videos and interactive content
* Use the tool to assess their personal HIV risk
* Receive support from trained peer educators (online)

The researchers hope this study will lead to new ways of using technology to improve HIV prevention and testing for young people.

DETAILED DESCRIPTION:
This study is designed to develop and evaluate a digital-based model for HIV education and self-screening aimed at increasing HIV-related knowledge, self-awareness of risk, and testing uptake among adolescents in Yogyakarta, Indonesia. Despite widespread access to digital technology, adolescent HIV testing coverage remains low due to stigma, limited knowledge, privacy concerns, and lack of youth-friendly services. The intervention model, named EKSTRIM (Edukasi dan Skrining HIV Mandiri), will be developed using a research and development framework based on the ADDIE model, which includes the stages of Analysis, Design, Development, Implementation, and Evaluation.

The study will proceed in three phases. In Phase I, an explanatory sequential mixed-methods design will be employed to assess the readiness, needs, and perceptions of adolescents and HIV program implementers regarding the use of digital platforms for HIV education and self-screening. Quantitative data will be collected through structured questionnaires, followed by qualitative data from focus group discussions and in-depth interviews. This phase will inform the technical and content requirements for the intervention.

Phase II will involve the design and development of the digital intervention model. The EKSTRIM platform will include interactive web-based modules on HIV prevention, a self-risk screening tool, peer educator support features, and links to adolescent-friendly HIV services. The platform will be evaluated using McCall's Quality Model to ensure functionality, reliability, and user-friendliness.

Phase III will test the effectiveness of the model using a double-blind, parallel-group randomized controlled trial with a pretest-posttest design. A total of 400 adolescents will be recruited using cluster random sampling from high schools in Yogyakarta. Participants will be randomly allocated to either the intervention group, which will access the EKSTRIM platform, or the control group, which will receive standard HIV educational materials. The intervention period will last six weeks.

Primary outcomes will include changes in HIV-related knowledge, self-awareness of HIV risk, and HIV testing uptake. Data analysis will involve general linear models, non-parametric tests (Wilcoxon and Mann-Whitney), difference-in-difference analysis, and multilevel linear modeling to assess the intervention's impact and identify contributing factors. It is anticipated that the digital intervention will lead to significant improvements in the targeted outcomes and that factors such as stigma, digital acceptance, and initial understanding of HIV will influence results.

This study aims to provide scientific evidence on the effectiveness of a digital, adolescent-centered HIV intervention that emphasizes privacy, peer support, and accessibility. The model is expected to be a scalable and sustainable solution for HIV prevention among youth and may inform broader policy and programmatic strategies at the local and national levels. Ethical approval will be obtained prior to study initiation, and all participants will provide informed consent or assent, with parental or guardian consent obtained as required under national regulations.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 15-17 years
* Reside or attend school in the Yogyakarta area
* Currently enrolled in one of the participating high schools
* Able to read and understand Bahasa Indonesia
* Own or have regular access to a smartphone or digital device with internet connectivity
* Provide informed assent to participate in the study
* Have obtained written parental or guardian consent

Exclusion Criteria:

* Adolescents outside the 15-17 age range
* Unable to access digital devices or internet independently
* Previously diagnosed with HIV (as this study targets prevention and self-screening among untested adolescents)
* Unwilling or unable to provide informed assent or whose parents/guardians do not provide consent
* Currently participating in another HIV-related intervention study

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV Testing Uptake Among Adolescents Using a Digital Self-Screening and Education Platform | Within 3 months after initial platform engagement
  Proportion of adolescents aged 15-17 who undergo voluntary HIV testing following engagement with the EKSTRIM digital platform, which includes audiovisual education, risk self-assessment, and online counseling. This outcome measures the effectiveness of the intervention in increasing HIV testing behavior compared to baseline where no participants had ever been tested, despite prior exposure to HIV-related information. Data will be collected through platform records and follow-up surveys to confirm testing uptake and linkage to services.

SECONDARY OUTCOMES:
Change in HIV Knowledge and Self Awareness Among Adolescents | From baseline to 4 weeks after initial platform use.
  Measured change in HIV-related knowledge and self-perceived risk awareness before and after using the EKSTRIM digital platform. Participants complete standardized pre- and post-intervention questionnaires assessing HIV transmission, prevention, testing, and risk awareness. The outcome evaluates the educational impact of audiovisual content and interactive modules. Scores will be compared using paired statistical analysis to determine knowledge gains and shifts in perceived vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: Rizka Ayu Setyani, Doctoral/PhD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Universitas Sebelas Maret, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and legal considerations related to adolescent privacy and consent. The study involves minors, and sharing of their sensitive health-related data, even in de-identified form, poses potential confidentiality risks. Data use is restricted by local institutional review board (IRB) protocols and national data protection regulations in Indonesia.

REFERENCES:
- [Background] Tang L, Wang J. Exploring the Relationship between Health Information Literacy and Health Behaviors of the Elderly. Iran J Public Health. 2023 Jul;52(7):1439-1446. doi: 10.18502/ijph.v52i7.13245. PMID 37593515
- [Background] Felsen UR, Tlamsa A, Moir L, Shukla S, Thompson D, Weiss JM, Heo M, Litwin AH. Comparing Routine HIV and Hepatitis C Virus Screening to Estimate the Effect of Required Consent on HIV Screening Rates Among Hospitalized Patients. Public Health Rep. 2022 Jan-Feb;137(1):102-109. doi: 10.1177/0033354921999170. Epub 2021 Mar 5. PMID 33673778
- [Background] Xiong S, Lu H, Peoples N, Duman EK, Najarro A, Ni Z, Gong E, Yin R, Ostbye T, Palileo-Villanueva LM, Doma R, Kafle S, Tian M, Yan LL. Digital health interventions for non-communicable disease management in primary health care in low-and middle-income countries. NPJ Digit Med. 2023 Feb 1;6(1):12. doi: 10.1038/s41746-023-00764-4. PMID 36725977
- [Background] Jenkins CL, Imran S, Mahmood A, Bradbury K, Murray E, Stevenson F, Hamilton FL. Digital Health Intervention Design and Deployment for Engaging Demographic Groups Likely to Be Affected by the Digital Divide: Protocol for a Systematic Scoping Review. JMIR Res Protoc. 2022 Mar 18;11(3):e32538. doi: 10.2196/32538. PMID 35302946
- [Background] Cheng AL, Leo AJ, Calfee RP, Dy CJ, Armbrecht MA, Abraham J. Multi-stakeholder perspectives regarding preferred modalities for mental health intervention delivered in the orthopedic clinic: a qualitative analysis. BMC Psychiatry. 2023 May 19;23(1):347. doi: 10.1186/s12888-023-04868-9. PMID 37208668
- [Background] Ibrahim MS, Mohamed Yusoff H, Abu Bakar YI, Thwe Aung MM, Abas MI, Ramli RA. Digital health for quality healthcare: A systematic mapping of review studies. Digit Health. 2022 Mar 18;8:20552076221085810. doi: 10.1177/20552076221085810. eCollection 2022 Jan-Dec. PMID 35340904
- [Background] Ninsiima M, Nyabigambo A, Kagaayi J. Acceptability of integration of cervical cancer screening into routine HIV care, associated factors and perceptions among HIV-infected women: a mixed methods study at Mbarara Regional Referral Hospital, Uganda. BMC Health Serv Res. 2023 Apr 3;23(1):333. doi: 10.1186/s12913-023-09326-6. PMID 37013535
- [Background] Putri WCWS, Ulandari LPS, Valerie IC, Prabowo BR, Hardiawan D, Sihaloho ED, Relaksana R, Wardhani BDK, Harjana NPA, Nugrahani NW, Siregar AYM, Januraga PP. Costs and scale-up costs of community-based Oral HIV Self-Testing for female sex workers and men who have sex with men in Jakarta and Bali, Indonesia. BMC Health Serv Res. 2024 Jan 22;24(1):114. doi: 10.1186/s12913-024-10577-0. PMID 38254186
- [Background] Johnston LG, Soe P, Widihastuti AS, Camellia A, Putri TA, Rakhmat FF, Nurwandani RA, Prabhu SM, Sulaiman N, Pronyk PM. Alarmingly High HIV Prevalence Among Adolescent and Young Men Who have Sex with Men (MSM) in Urban Indonesia. AIDS Behav. 2021 Nov;25(11):3687-3694. doi: 10.1007/s10461-021-03347-0. Epub 2021 Jun 18. PMID 34143341
- [Background] Yoon J, Lee M, Ahn JS, Oh D, Shin SY, Chang YJ, Cho J. Development and Validation of Digital Health Technology Literacy Assessment Questionnaire. J Med Syst. 2022 Jan 24;46(2):13. doi: 10.1007/s10916-022-01800-8. PMID 35072816
- See also: EKSTRIM study protocol — https://drive.google.com/file/d/18K8ImooxCYP9CJ7Vpxg1NBH6ySyYy1Tr/view?usp=sharing
- Available data/document: Study Protocol: EKSTRIM study protocol — https://drive.google.com/file/d/18K8ImooxCYP9CJ7Vpxg1NBH6ySyYy1Tr/view?usp=sharing — This study does not plan to share individual participant data (IPD) due to the involvement of minors and the sensitive nature of HIV-related information. The protocol prioritizes adolescent privacy, confidentiality, and protection of digital health data in accordance with national regulations and institutional ethical standards. Sharing of IPD, even in de-identified form, may risk re-identification, especially in small or specific community samples. All collected data will be stored securely and accessed only by authorized study personnel. Aggregated results may be shared in publications and presentations, but raw IPD will remain confidential.
- Available data/document: Informed Consent Form: EKSTRIM_ICF — https://drive.google.com/file/d/1cnEfDqkpzy54F8jV8atQ161KA-9C9gwW/view?usp=sharing — The EKSTRIM Informed Consent Form is clearly structured and comprehensive, addressing all essential components of ethical research. It outlines the study's objectives, procedures, risks, benefits, and rights of participants in a language that is accessible and age-appropriate for adolescents. It emphasizes voluntary participation and the right to withdraw at any time without consequence. The form includes detailed information on data confidentiality, compensation, and peer educator support, enhancing participant protection and engagement. The inclusion of contact information offers transparency and accessibility. However, the form could be strengthened by explicitly stating how long data will be retained and whether participants will receive feedback on study findings. Overall, the ICF demonstrates ethical rigor and appropriateness for adolescent involvement in HIV-related digital health research.